CLINICAL TRIAL: NCT02045992
Title: Effect of High-dose Caffeine on Cardiac Arrhythmias in Patients With Heart Failure - a Randomized Clinical Trial
Brief Title: Arrhythmic Effects of Hight Dose Caffeine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luis Eduardo Paim Rohde (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Luis Eduardo Paim Rohde, Professor, Hospital de Clinicas de Porto Alegre
Organization: Hospital de Clinicas de Porto Alegre (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 110298
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine (Experimental): Caffeine 500mg
  Interventions: Dietary Supplement: caffeine
- Placebo (Placebo Comparator): Lactose 500mg

INTERVENTIONS:
Dietary Supplement: caffeine — Five doses of 100mg of caffeine diluted in 100 ml of decaffeinated coffee. One dose every hour for five hours
  Arms: Caffeine

SUMMARY:
Heart failure patients represent a group of individuals at higher risk for cardiac arrhythmias. There is a perception that caffeine consumption may represent an increase in this risk. Although the medical staff and health professionals suggest a reduction in the intake of this substance to patients considered at risk, there is no scientific proof for this recommendation.

Some animal studies suggest a possible association between arrhythmias and caffeine use with higher doses, but this finding did not appear in human studies. In particular, little is known about the association between caffeine consumption and arrhythmias in patients with heart failure, especially at higher doses of consumption.

More specific and safe guidelines on caffeine consumption are needed.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure in NYHA functional class I-III
* LV Ejection fraction <45%
* Age > 18 y.o.
* Cardio-defibrillator implanted with normal functioning with at least 30 days.

Exclusion Criteria:

* Impossibility of take caffeine
* Inability to perform an exercise test
* Initial use of amiodarone in the last 2 months
* Unstable ventricular arrhythmias, shock or ATP in the last 60 days
* Hospitalization in the last two months due to decompensated heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Arrhythmias | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Zuchinali P, Souza GC, Pimentel M, Chemello D, Zimerman A, Giaretta V, Salamoni J, Fracasso B, Zimerman LI, Rohde LE. Short-term Effects of High-Dose Caffeine on Cardiac Arrhythmias in Patients With Heart Failure: A Randomized Clinical Trial. JAMA Intern Med. 2016 Dec 1;176(12):1752-1759. doi: 10.1001/jamainternmed.2016.6374. PMID 27749954